CLINICAL TRIAL: NCT02975271
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Tolerability of Serlopitant for the Treatment of Pruritus Following Burn Injury
Brief Title: Study of the Efficacy, Safety & Tolerability of Serlopitant for Pruritus (Itch) After Burn Injury
Acronym: AUBURN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTI-104
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Pruritus; Burns
MeSH Terms: conditions — Pruritus; Burns | interventions — serlopitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Serlopitant (Experimental): Dose of experimental drug Serlopitant
  Interventions: Drug: Serlopitant
- Placebo (Placebo Comparator): Matching dose of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Serlopitant
  Arms: Serlopitant
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
Study of the Efficacy, Safety & Tolerability of Serlopitant for Pruritus (Itch) After Burn Injury

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, age 18-65 years at consent.
* History of serious burn injury
* Pruritus (itchiness) prior to the initial screening visit and during the screening period
* Judged to be in good health in the investigator's opinion.

Key Exclusion Criteria:

* Prior treatment with study drug or similar drug
* Pruritus (itchiness) due to another reason besides burn injury/ healing.
* Presence of any medical condition or disability that, in the investigator's opinion, could interfere with the assessment of safety or efficacy in this trial or compromise the safety of the subject.
* History of hypersensitivity to study drug or any of its components.
* Currently pregnant or male partner of pregnant female.
* Females of childbearing potential who are unable or unwilling to use adequate contraception or who are breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Change in Itch Intensity - Numeric Rating Scale | Week 6

SECONDARY OUTCOMES:
Itch Intensity Responder Rate - Numeric Rating Scale | Week 6

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Study Site 404, Phoenix, Arizona
  - Study Site 402, Washington D.C., District of Columbia
  - Study Site 412, Gainesville, Florida
  - Study Site 403, Tampa, Florida
  - Study Site 409, Lincoln, Nebraska
  - Study Site 401, Winston-Salem, North Carolina
  - Study Site 413, Seattle, Washington